CLINICAL TRIAL: NCT06491927
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of RGX-202 Gene Therapy in Males With Duchenne Muscular Dystrophy (DMD)
Brief Title: Long Term Follow-up for RGX-202
Status: Enrolling by invitation | Type: Observational
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-202-5101
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Gene therapy; DMD; Duchenne; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RGX-202 Recipients: Subjects who have received RGX-202 in a separate parent study.
  Interventions: Genetic: No Intervention

INTERVENTIONS:
Genetic: No Intervention — Observational study

SUMMARY:
RGX-202-5101 is a long-term follow up study that evaluates the long term safety and efficacy of RGX-202 in participants who have received RGX-202 (a gene therapy designed to deliver a transgene for novel microdystrophin that includes functional elements of naturally-occurring dystrophin including the C-Terminal (CT) domain) in a separate parent study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational study to evaluate the long-term safety and efficacy of RGX-202. Eligible participants are those who have undergone evaluation in a previous (parent) clinical study following a single intravenous infusion of RGX-202 for the treatment of DMD. Enrollment in the current long-term follow-up (LTFU) study will occur after the participant has completed or discontinued from the parent study. Participants will be followed in this study cumulatively for up to 5 years after RGX-202 administration (inclusive of the parent study). No investigational treatment will be administered under this protocol. The total study duration for each participant may vary depending on when he enrolls in the current study following RGX-202 administration in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* The parent(s) or legal guardian(s) of the participant has/(have) provided written informed consent and (where applicable) Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been explained, prior to any research-related procedures; and, where applicable, the minor participant has provided written or verbal assent according to local requirements.
* Must have undergone evaluation in a previous clinical study following a single IV infusion of RGX-202 for the treatment of DMD and either completed or withdrawn early from that study.
* Participant and parent(s)/legal guardian(s) are willing and able to comply with scheduled visits, and study procedures.
* Sexually active participants must be willing to use a medically accepted method of contraception from the time of the screening visit through 5 years after RGX-202 administration.

Exclusion Criteria:

* No exclusion criteria apply in this observational follow up study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Received RGX-202 in a separate parent study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of long-term safety of RGX-202 | 5 years inclusive of parent study
  Incidences of AEs and SAEs over time

SECONDARY OUTCOMES:
Efficacy measured by change in Functional Assessment | 5 years inclusive of parent study
  Longitudinal trajectory (mean and change from baseline) in North Star Ambulatory Assessment (NSAA) raw and linear score

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois